CLINICAL TRIAL: NCT06067139
Title: Sleep for Health: A Randomized Clinical Trial Examining the Effects of Cognitive Behavioral Therapy for Insomnia on Diabetes Risk
Brief Title: Sleep for Health Study on the Effects of Cognitive Behavioral Therapy for Insomnia on Diabetes Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DK132229 (NIH); 1R01DK132229-01A1 (NIH)
Record Dates: First submitted 2023-07-31; First posted 2023-10-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 2; Prediabetic State; Sleep Initiation and Maintenance Disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital cognitive behavioral therapy (dCBT-I) (Experimental): CBT-I is designed to change sleep habits and scheduling factors that affect sleep, and to address misconceptions about sleep and insomnia that perpetuate sleep difficulties. The investigators will employ SHUTi, which is an extensively studied dCBT-I program. SHUTi is intended to improve insomnia symptoms by providing neurobehavioral intervention (cognitive behavioral therapy for insomnia - CBT-I) in adults with chronic insomnia. It is a six-core internet-delivered CBT-I web-based app that is run through a browser. It is accessible via iPhone/iPad, Android phone/tablet, computer or laptop (any device with a browser). SHUTi follows evidence-based CBT-I principles.
  Interventions: Other: SHUTi
- Patient Education (PE) (Active Comparator): Participants will be given access to a patient education website. It will provide nontailored material about insomnia symptoms; the impact, prevalence, and causes of insomnia; and basic lifestyle, environmental, and behavioral strategies to improve sleep.
  Interventions: Other: Patient Education

INTERVENTIONS:
Other: SHUTi — Each core includes a variety of interactive features, such as animations, vignettes, "myth" and "reality" buttons that reveal common misperceptions and facts about sleep, "learn more" buttons that provide in-depth information about a topic, and quizzes. All cores follow a similar structure with objectives, main content, homework, and review. Participants are free to revisit cores as many times as they like.
  Arms: Digital cognitive behavioral therapy (dCBT-I)
Other: Patient Education — The PE website will present content in a simple, static form, without interactive components; and all content on the website will be provided at once, rather than in modules that unlock over time. The PE website will also not provide personalized or individually tailored treatment recommendations.
  Arms: Patient Education (PE)

SUMMARY:
This study tests whether providing cognitive behavioral therapy for insomnia (CBT-I) to people with prediabetes results in a reduction in glucose levels compared to a patient education control program.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2D) is a major cause of blindness, kidney failure, cardiovascular disease, amputations, reduced quality of life, and premature death in the United States, and it is expected that one in three Americans will have T2D by 2050. To stem the tide of this health crisis, new strategies are needed to prevent the progression to T2D from prediabetes-elevated glucose levels that are not yet in the diabetes range. A growing body of research suggests that insomnia is a major modifiable risk factor for progression to diabetes. The proposed study would build off a promising feasibility study to test whether providing cognitive behavioral therapy for insomnia (CBT-I) to patients with prediabetes results in a reduction in glucose levels compared to a patient education control program. If so, this insomnia treatment could be an effective tool to prevent diabetes.

Individuals with prediabetes and insomnia will be randomized to receive six sessions of a deployment-ready digital CBT-I program, providing standard-of-care treatment for insomnia (intervention arm, n = 150), or a patient education website providing nontailored material about insomnia (control arm, n = 150). The investigators will complete assessments at baseline, at 11 weeks (after the conclusion of the intervention and control programs), and at 33 weeks post-baseline, measuring hyperglycemia, objective and subjective measures of sleep, and potential mediating variables including diet, exercise, and mood.

The investigators will assess (1) whether individuals randomized to the intervention arm have lower rates of hyperglycemia, as measured by oral glucose tolerance testing and various secondary measures, than individuals randomized to the control arm at 11 weeks and 33 weeks after baseline; (2) whether improvements in sleep after baseline are associated with decreases in hyperglycemia, regardless of study arm; and (3) whether any effects of the intervention on hyperglycemia are mediated by improvements in sleep, diet, exercise, and/or mood.

This research will serve as a critical step in identifying a potentially dramatic tool for improving health outcomes for Americans at risk of T2DM. Sleep interventions can lead to sustained improvements that are intrinsically rewarding to patients. If effective, digital CBT-I could provide a powerful pathway to preventing diabetes for millions of patients with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years and < 80 years of age
* Prediabetes
* Insomnia
* Regular access to device with internet access
* Adequate data at baseline

Exclusion Criteria:

* BMI > 40 kg/m2
* Sleep comorbidities detected in medical record or via medical history
* Shift work or significant, externally imposed irregular sleep schedule
* moderate to severe OSA by home sleep apnea test as part of trial protocol
* Received a full course of CBT-I in the last 12 months
* Current use of medication with glycemic effects:
* History of type 1 or type 2 diabetes or recent/planned use of hypoglycemic agents (e.g., metformin, insulin)
* Recent history of bariatric surgery or planning bariatric surgery in the next year
* Current or recent use of weight loss meds
* Unstable sleep medication regimen (recent change to schedule or dosage)
* Significant comorbidity that may interfere with CBT-I uptake or increase risks
* Unwilling or unable to limit heavy machinery use/long bouts of driving or unstable illness that would be worsened by sleep restriction
* High risk of falls
* Epilepsy
* Medical conditions that interfere with dCBT-I or contribute to insomnia or diabetes risk (e.g., hyperthyroidism, significant kidney disease, active cancer treatment, any medical condition that requires chronic steroid use)
* Significant alcohol or substance use disorder
* Active or recent history of eating disorder, recent weight change of >10%
* Women: pregnancy (current or planned), breastfeeding, < 1 year postpartum
* Use of hydroxyurea
* Extensive skin changes or adhesive allergy making CGM sensor use problematic

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
2-hour post-load glucose (2hPG) (mg/dL) | V1 (baseline), V2 (11 weeks after randomization), V3 (33 weeks from randomization)
  2-hour post-load glucose (mg/dL)

SECONDARY OUTCOMES:
Hemoglobin A1c (A1C) (percentage) | V1 (baseline), V2 (11 weeks after randomization), V3 (33 weeks from randomization)
  Plasma HgB A1C (percentage)
Fasting plasma glucose (FPG) (mg/dL) | V1 (baseline), V2 (11 weeks after randomization), V3 (33 weeks from randomization)
  Fasting plasma glucose levels (mg/dL)
Mean glucose on CGM (mg/dL) | V1 (baseline), V2 (11 weeks after randomization), V3 (33 weeks from randomization)
  Average blood glucose levels throughout CGM wear duration (mg/dL)
Insulin resistance score (probability ranking, Calculated using the insulin and C-peptide concentrations converted to pmol/L) | V1 (baseline), V2 (11 weeks after randomization), V3 (33 weeks from randomization)
  Insulin resistance score - (probability ranking, Calculated using the insulin and C-peptide concentrations converted to pmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Erin LeBlanc, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers after the end of the study.

REFERENCES:
- [Background] Tabak AG, Herder C, Rathmann W, Brunner EJ, Kivimaki M. Prediabetes: a high-risk state for diabetes development. Lancet. 2012 Jun 16;379(9833):2279-90. doi: 10.1016/S0140-6736(12)60283-9. Epub 2012 Jun 9. PMID 22683128
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Centers for Disease Control and Prevention. Diabetes Report Card 2014. Atlanta, GA: Centers for Disease Control and Prevention, US Dept of Health and Human Services, 2015.
- [Background] LeBlanc ES, Smith NX, Nichols GA, Allison MJ, Clarke GN. Insomnia is associated with an increased risk of type 2 diabetes in the clinical setting. BMJ Open Diabetes Res Care. 2018 Dec 26;6(1):e000604. doi: 10.1136/bmjdrc-2018-000604. eCollection 2018. PMID 30687505
- [Background] Anothaisintawee T, Reutrakul S, Van Cauter E, Thakkinstian A. Sleep disturbances compared to traditional risk factors for diabetes development: Systematic review and meta-analysis. Sleep Med Rev. 2016 Dec;30:11-24. doi: 10.1016/j.smrv.2015.10.002. Epub 2015 Oct 21. PMID 26687279
- [Background] Cappuccio FP, D'Elia L, Strazzullo P, Miller MA. Quantity and quality of sleep and incidence of type 2 diabetes: a systematic review and meta-analysis. Diabetes Care. 2010 Feb;33(2):414-20. doi: 10.2337/dc09-1124. Epub 2009 Nov 12. PMID 19910503
- [Background] Hatoum HT, Kania CM, Kong SX, Wong JM, Mendelson WB. Prevalence of insomnia: a survey of the enrollees at five managed care organizations. Am J Manag Care. 1998 Jan;4(1):79-86. PMID 10179908
- [Background] Spiegel K, Leproult R, Van Cauter E. Impact of sleep debt on metabolic and endocrine function. Lancet. 1999 Oct 23;354(9188):1435-9. doi: 10.1016/S0140-6736(99)01376-8. PMID 10543671
- [Background] van Leeuwen WM, Hublin C, Sallinen M, Harma M, Hirvonen A, Porkka-Heiskanen T. Prolonged sleep restriction affects glucose metabolism in healthy young men. Int J Endocrinol. 2010;2010:108641. doi: 10.1155/2010/108641. Epub 2010 Apr 19. PMID 20414467
- [Background] Leproult R, Holmback U, Van Cauter E. Circadian misalignment augments markers of insulin resistance and inflammation, independently of sleep loss. Diabetes. 2014 Jun;63(6):1860-9. doi: 10.2337/db13-1546. Epub 2014 Jan 23. PMID 24458353
- [Background] Stamatakis KA, Punjabi NM. Effects of sleep fragmentation on glucose metabolism in normal subjects. Chest. 2010 Jan;137(1):95-101. doi: 10.1378/chest.09-0791. Epub 2009 Jun 19. PMID 19542260
- [Background] Buxton OM, Pavlova M, Reid EW, Wang W, Simonson DC, Adler GK. Sleep restriction for 1 week reduces insulin sensitivity in healthy men. Diabetes. 2010 Sep;59(9):2126-33. doi: 10.2337/db09-0699. Epub 2010 Jun 28. PMID 20585000
- [Background] Gale JE, Cox HI, Qian J, Block GD, Colwell CS, Matveyenko AV. Disruption of circadian rhythms accelerates development of diabetes through pancreatic beta-cell loss and dysfunction. J Biol Rhythms. 2011 Oct;26(5):423-33. doi: 10.1177/0748730411416341. PMID 21921296
- [Background] Nedeltcheva AV, Kilkus JM, Imperial J, Kasza K, Schoeller DA, Penev PD. Sleep curtailment is accompanied by increased intake of calories from snacks. Am J Clin Nutr. 2009 Jan;89(1):126-33. doi: 10.3945/ajcn.2008.26574. Epub 2008 Dec 3. PMID 19056602
- [Background] Patel SR, Hu FB. Short sleep duration and weight gain: a systematic review. Obesity (Silver Spring). 2008 Mar;16(3):643-53. doi: 10.1038/oby.2007.118. Epub 2008 Jan 17. PMID 18239586
- [Background] Patel SR. Reduced sleep as an obesity risk factor. Obes Rev. 2009 Nov;10 Suppl 2:61-8. doi: 10.1111/j.1467-789X.2009.00664.x. PMID 19849803
- [Background] Patel SR, Blackwell T, Redline S, Ancoli-Israel S, Cauley JA, Hillier TA, Lewis CE, Orwoll ES, Stefanick ML, Taylor BC, Yaffe K, Stone KL; Osteoporotic Fractures in Men Research Group; Study of Osteoporotic Fractures Research Group. The association between sleep duration and obesity in older adults. Int J Obes (Lond). 2008 Dec;32(12):1825-34. doi: 10.1038/ijo.2008.198. Epub 2008 Oct 21. PMID 18936766
- [Background] Booth JN, Bromley LE, Darukhanavala AP, Whitmore HR, Imperial JG, Penev PD. Reduced physical activity in adults at risk for type 2 diabetes who curtail their sleep. Obesity (Silver Spring). 2012 Feb;20(2):278-84. doi: 10.1038/oby.2011.306. Epub 2011 Oct 13. PMID 21996665
- [Background] Broussard JL, Wroblewski K, Kilkus JM, Tasali E. Two Nights of Recovery Sleep Reverses the Effects of Short-term Sleep Restriction on Diabetes Risk. Diabetes Care. 2016 Mar;39(3):e40-1. doi: 10.2337/dc15-2214. Epub 2016 Jan 19. No abstract available. PMID 26786578
- [Background] Thiesse L, Rudzik F, Spiegel K, Leproult R, Pieren R, Wunderli JM, Foraster M, Heritier H, Eze IC, Meyer M, Vienneau D, Brink M, Probst-Hensch N, Roosli M, Cajochen C. Adverse impact of nocturnal transportation noise on glucose regulation in healthy young adults: Effect of different noise scenarios. Environ Int. 2018 Dec;121(Pt 1):1011-1023. doi: 10.1016/j.envint.2018.05.036. Epub 2018 Jul 4. PMID 30408889
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Cho YW, Kim KT, Moon HJ, Korostyshevskiy VR, Motamedi GK, Yang KI. Comorbid Insomnia With Obstructive Sleep Apnea: Clinical Characteristics and Risk Factors. J Clin Sleep Med. 2018 Mar 15;14(3):409-417. doi: 10.5664/jcsm.6988. PMID 29458695
- [Background] American Diabetes Association. 3. Prevention or Delay of Type 2 Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S34-S39. doi: 10.2337/dc21-S003. PMID 33298414
- [Background] Asarnow JR, Jaycox LH, Duan N, LaBorde AP, Rea MM, Murray P, Anderson M, Landon C, Tang L, Wells KB. Effectiveness of a quality improvement intervention for adolescent depression in primary care clinics: a randomized controlled trial. JAMA. 2005 Jan 19;293(3):311-9. doi: 10.1001/jama.293.3.311. PMID 15657324
- [Background] The Diabetes Prevention Program Research Group. The Diabetes Prevention Program: baseline characteristics of the randomized cohort. The Diabetes Prevention Program Research Group. Diabetes Care. 2000 Nov;23(11):1619-29. doi: 10.2337/diacare.23.11.1619. PMID 11092283
- [Background] Nedeltcheva AV, Kessler L, Imperial J, Penev PD. Exposure to recurrent sleep restriction in the setting of high caloric intake and physical inactivity results in increased insulin resistance and reduced glucose tolerance. J Clin Endocrinol Metab. 2009 Sep;94(9):3242-50. doi: 10.1210/jc.2009-0483. Epub 2009 Jun 30. PMID 19567526
- [Background] Lindstrom J, Louheranta A, Mannelin M, Rastas M, Salminen V, Eriksson J, Uusitupa M, Tuomilehto J; Finnish Diabetes Prevention Study Group. The Finnish Diabetes Prevention Study (DPS): Lifestyle intervention and 3-year results on diet and physical activity. Diabetes Care. 2003 Dec;26(12):3230-6. doi: 10.2337/diacare.26.12.3230. PMID 14633807
- [Background] Kothari V, Cardona Z, Chirakalwasan N, Anothaisintawee T, Reutrakul S. Sleep interventions and glucose metabolism: systematic review and meta-analysis. Sleep Med. 2021 Feb;78:24-35. doi: 10.1016/j.sleep.2020.11.035. Epub 2020 Dec 7. PMID 33383394
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Hanefeld M, Sulk S, Helbig M, Thomas A, Kohler C. Differences in Glycemic Variability Between Normoglycemic and Prediabetic Subjects. J Diabetes Sci Technol. 2014 Mar;8(2):286-290. doi: 10.1177/1932296814522739. Epub 2014 Mar 2. PMID 24876580
- [Background] Cohen J. Statistical Power Analysis for the Behavioral Sciences. 2nd ed: Lawrence Erlbaum Associates; 1988.
- [Background] Rubin DB. Multiple Imputation for Nonresponse in Surveys. New York: John Wiley & Sons, Inc.; 1987.
- [Background] Krishnan V, Collop NA. Gender differences in sleep disorders. Curr Opin Pulm Med. 2006 Nov;12(6):383-9. doi: 10.1097/01.mcp.0000245705.69440.6a. PMID 17053485
- [Background] Nosek BA, Spies JR, Motyl M. Scientific Utopia: II. Restructuring Incentives and Practices to Promote Truth Over Publishability. Perspect Psychol Sci. 2012 Nov;7(6):615-31. doi: 10.1177/1745691612459058. PMID 26168121
- [Derived] LeBlanc ES, Smith N, Hwang D, Young DR, Oshiro C, Mayhew M, Massimino S, Catlin C, Clarke G. The sleep for health study: A randomized clinical trial of the impact of insomnia treatment on glycemia in people with prediabetes. Contemp Clin Trials. 2025 Feb;149:107796. doi: 10.1016/j.cct.2024.107796. Epub 2024 Dec 25. PMID 39730078
- See also: Diabetes Care and Education Dietetic Practice Group. What is pre-diabetes? — http://dbcms.s3.amazonaws.com/media/files/80cc1018-d357-49de-91df-2bd298499dc2/what%20is%20prediabetes.pdf
- See also: American Diabetes Association. All about pre-diabetes. Toolkit No. 3 2012 — http://professional.diabetes.org/
- See also: Dexcom G6 Pro — https://provider.dexcom.com/faqs-categories/dexcom-g6-pro